CLINICAL TRIAL: NCT06091982
Title: The Need of Renal Replacement Therapy and In-Hospital Mortality Incidence In Patients With Cardiac Surgery Associated Acute Kidney Injury: Retrospective Study
Brief Title: Renal Replacement Therapy and In-Hospital Mortality Incidence in Cardiac Surgery Associated Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Prieta Adriane MD, MD Anesthesiologist, National Cardiovascular Center Harapan Kita Hospital Indonesia
Other Study IDs: 01.202308.101
Record Dates: First submitted 2023-10-08; First posted 2023-10-23 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury (AKI); Cardiac Surgery; Renal Replacement Therapy; Mortality
MeSH Terms: conditions — Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI-RRT: Post cardiovascular surgery patients with condition of acute kidney injury postoperative; and with an exposure of renal replacement therapy (intermittent haemodialysis or continuous renal replacement therapy) which is indicated postoperatively.
  Interventions: Procedure: Renal Replacement Therapy (RRT)
- AKI non RRT: Post cardiovascular surgery patients with condition of acute kidney injury postoperative; but without exposure of renal replacement therapy.

INTERVENTIONS:
Procedure: Renal Replacement Therapy (RRT) — Renal Support therapy which consist of procedure of intermittent hemodialysis (IHD) or continuous veno-venous hemofiltration/hemodialysis/hemodiafiltration (CVVH/CVVHD/CVVHDF)
  Groups: AKI-RRT

SUMMARY:
The goal of this study is to analyse the relation of severe acute kidney injury post cardiac surgery which characterised by the need of renal replacement therapy, with in-hospital postoperative mortality incidence.

The main question it aims to answer:

To compare between patients complicated with acute kidney injury and exposure of renal replacement therapy (AKI-RRT) and patients complicated with acute kidney injury which does not require renal replacement therapy, in associated with in-hospital postoperative mortality.

DETAILED DESCRIPTION:
Type of study: observational study

Participant population: Post cardiac surgery patients with condition of acute kidney injury postoperative, will be assigned into 2 groups, based on their exposure to renal replacement therapy. Those groups are:

Group AKI-RRT : patients with AKI postoperative with exposure of renal replacement therapy Group AKI non RRT : patients with AKI postoperative, with no exposure to renal replacement therapy Researchers will compare group AKI-RRT and AKI non RRT to analyse the association to postoperative mortality, and other factors that related to mortality variable.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are at least 18 years old, underwent cardiac surgery in Harapan Kita National Cardiovascular Center from January 2020 to December 2022.
2. Patients with condition was complicated with Acute Kidney Injury (AKI) which was characterised by an increase in serum creatinine > 0.3 mg/dL or > 150% of the preoperative serum creatinine value, which was checked within 12 hours post-operative.
3. All patients' data is recorded in the medical records unit.

Exclusion Criteria:

1. Patients with previous history of dialysis or renal failure in dialysis.
2. Incomplete or loss of patients' data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients with condition of acute kidney injury postoperative, which underwent the surgery from January 2020 to December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1113 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Widyantoro, PhD, Study Chair — Institutional Review Board
Locations (1):
- National Cardiovascular Center, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yi Q, Li K, Jian Z, Xiao YB, Chen L, Zhang Y, Ma RY. Risk Factors for Acute Kidney Injury after Cardiovascular Surgery: Evidence from 2,157 Cases and 49,777 Controls - A Meta-Analysis. Cardiorenal Med. 2016 May;6(3):237-50. doi: 10.1159/000444094. Epub 2016 Mar 17. PMID 27275160
- [Background] Thakar CV, Arrigain S, Worley S, Yared JP, Paganini EP. A clinical score to predict acute renal failure after cardiac surgery. J Am Soc Nephrol. 2005 Jan;16(1):162-8. doi: 10.1681/ASN.2004040331. Epub 2004 Nov 24. PMID 15563569
- [Background] Vives M, Hernandez A, Parramon F, Estanyol N, Pardina B, Munoz A, Alvarez P, Hernandez C. Acute kidney injury after cardiac surgery: prevalence, impact and management challenges. Int J Nephrol Renovasc Dis. 2019 Jul 2;12:153-166. doi: 10.2147/IJNRD.S167477. eCollection 2019. PMID 31303781
- [Background] Olivero JJ, Olivero JJ, Nguyen PT, Kagan A. Acute kidney injury after cardiovascular surgery: an overview. Methodist Debakey Cardiovasc J. 2012 Jul-Sep;8(3):31-6. doi: 10.14797/mdcj-8-3-31. PMID 23227284
- [Background] Carrascal Y, Laguna G, Blanco M, Paneda L, Segura B. Acute Kidney Injury after Heart Valve Surgery in Elderly Patients: any Risk Factors to Modify? Braz J Cardiovasc Surg. 2021 Feb 1;36(1):1-9. doi: 10.21470/1678-9741-2019-0483. PMID 33113315
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Bove T, Calabro MG, Landoni G, Aletti G, Marino G, Crescenzi G, Rosica C, Zangrillo A. The incidence and risk of acute renal failure after cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Aug;18(4):442-5. doi: 10.1053/j.jvca.2004.05.021. PMID 15365924
- [Background] Liu C, Zhang HT, Yue LJ, Li ZS, Pan K, Chen Z, Gu SP, Pan T, Pan J, Wang DJ. Risk factors for mortality in patients undergoing continuous renal replacement therapy after cardiac surgery. BMC Cardiovasc Disord. 2021 Oct 21;21(1):509. doi: 10.1186/s12872-021-02324-8. PMID 34674651
- [Background] Oh TK, Song IA. Postoperative acute kidney injury requiring continuous renal replacement therapy and outcomes after coronary artery bypass grafting: a nationwide cohort study. J Cardiothorac Surg. 2021 Oct 26;16(1):315. doi: 10.1186/s13019-021-01704-7. PMID 34702324
- [Background] Zou H, Hong Q, Xu G. Early versus late initiation of renal replacement therapy impacts mortality in patients with acute kidney injury post cardiac surgery: a meta-analysis. Crit Care. 2017 Jun 17;21(1):150. doi: 10.1186/s13054-017-1707-0. PMID 28623953
- [Background] Borisov AS, Malov AA, Kolesnikov SV, Lomivorotov VV. Renal Replacement Therapy in Adult Patients After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Aug;33(8):2273-2286. doi: 10.1053/j.jvca.2019.02.023. Epub 2019 Feb 15. No abstract available. PMID 30871949
- [Background] Matsuura R, Iwagami M, Moriya H, Ohtake T, Hamasaki Y, Nangaku M, Doi K, Kobayashi S, Noiri E. The Clinical Course of Acute Kidney Disease after Cardiac Surgery: A Retrospective Observational Study. Sci Rep. 2020 Apr 16;10(1):6490. doi: 10.1038/s41598-020-62981-1. PMID 32300140
- [Background] Thongprayoon C, Cheungpasitporn W, Shah IK, Kashyap R, Park SJ, Kashani K, Dillon JJ. Long-term Outcomes and Prognostic Factors for Patients Requiring Renal Replacement Therapy After Cardiac Surgery. Mayo Clin Proc. 2015 Jul;90(7):857-64. doi: 10.1016/j.mayocp.2015.03.026. PMID 26141328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all adult cardiac surgery patients (> 18 years old) with EMRs who were admitted to the cardiac surgery ICU from January 1st , 2020 to December 31st, 2022
Pre-assignment Details: 2.670 patients excluded due to incomplete/missing reports/data, with previous RRT before surgery, and not complicated with CSA-AKI
Period: Overall Study
Arm/Group | AKI-RRT | AKI Non RRT
Started | 302 | 811
Completed | 302 | 811
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subject number: people
Groups:
- AKI RRT: Post cardiovascular surgery patients with condition of acute kidney injury postoperative; and with an exposure of renal replacement therapy (intermittent haemodialysis or continuous renal replacement therapy) which is indicated postoperatively.
- Total: Total of all reporting groups
Arm/Group | AKI RRT | AKI Non RRT | Total
Number analyzed (Participants) | 302 | 811 | 1113
Age, Customized [Count of Participants; unit: Participants] — Subject's age by the time of surgery, whose aged > 60 years old
  Participants
    > 60 years old | 196 | 219 | 415
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 170 | 251
  Male | 221 | 641 | 862
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Surgery [Count of Participants; unit: Participants] — Number of participants in one type of surgery
  Participants
    CABG | 118 | 425 | 543
    Valves | 83 | 216 | 299
    Mixed Valves | 38 | 66 | 104
    Congenital | 14 | 39 | 53
    Other surgeries | 49 | 65 | 114
Diabetes [Count of Participants; unit: Participants] — Number of participants who had diabetes history
  Participants | 121 | 240 | 361
Hypertension [Count of Participants; unit: Participants] — Number of participant who had hypertensive disease
  Participants | 118 | 315 | 433
History of stroke [Count of Participants; unit: Participants] — Number of participants with history of stroke
  Participants | 118 | 315 | 433
Smoker [Count of Participants; unit: Participants] — Number of participant who is currently a smoker
  Participants | 62 | 132 | 194
Renal disease [Count of Participants; unit: Participants] — Number of participant which has a renal disease
  Participants | 10 | 7 | 17
Creatinine level > 3.0 mg/dL [Count of Participants; unit: Participants] — Number of participant with creatinine level postoperative more than 3.0 gr/dL
  Participants | 81 | 51 | 132
Use of inotropes and vasoactives > 2 drugs [Count of Participants; unit: Participants] — Number of participants who required inotrope and/or vasoactive drugs more than 2 kinds.
  Participants | 129 | 151 | 280
Postoperative diuretic therapy [Count of Participants; unit: Participants] — Number of participants who required diuretic therapy postoperative
  Participants | 217 | 590 | 807

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of participants who died of any cause during postoperative care in hospital
Time Frame: From ICU admission postoperative until the death date during hospital care, assessed up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | AKI-RRT | AKI Non RRT
Number analyzed (Participants) | 302 | 811
Participants | 96 | 34
Statistical Analysis 1: Comparison: AKI-RRT vs AKI Non RRT; Bivariable analysis of both groups; Test type: Superiority; p < 0.0001, Chi-squared; Odds Ratio (OR) = 10.6, 95% CI 2-sided [7.0 to 16.2]
Statistical Analysis 2: Comparison: AKI-RRT; Multivariable analysis; Test type: Other — Multiple logistic regression; p < 0.0001, Regression, Logistic; Odds Ratio, log = 3.4, 95% CI 2-sided [2.0 to 6.1]

2. Secondary Outcome: ICU Stay Over 5 Days
Description: Number of participants which the postoperative ICU length of stay more than 5 days
Time Frame: Time of ICU length of stay measured with days, up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AKI-RRT | AKI Non RRT
Number analyzed (Participants) | 302 | 811
Participants | 183 | 89
Statistical Analysis 1: Comparison: AKI-RRT vs AKI Non RRT; Test type: Superiority; p < 0.0001, Chi-squared; Odds Ratio (OR) = 12.5, 95% CI 2-sided [9.1 to 17.1]
Statistical Analysis 2: Comparison: AKI-RRT; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio, log = 4.4, 95% CI 2-sided [2.8 to 7.0]

3. Secondary Outcome: Mechanical Ventilation > 48 Hours
Description: Number of participants which the postoperative usage of mechanical ventilation (breathing ventilator) more than 48 hours
Time Frame: Time of ventilator usage measure with hours, up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AKI-RRT | AKI Non RRT
Number analyzed (Participants) | 302 | 811
Participants | 198 | 88
Statistical Analysis 1: Comparison: AKI-RRT vs AKI Non RRT; Test type: Superiority; p < 0.0001, Chi-squared; Odds Ratio (OR) = 15.6, 95% CI 2-sided [11.3 to 21.6]
Statistical Analysis 2: Comparison: AKI-RRT; Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio, log = 5.2, 95% CI 2-sided [3.3 to 8.2]

ADVERSE EVENTS:
Time Frame: Adverse events that occurred from postoperative period until 1 month after discharged based on electronic medical records
Description: Any additional diagnosis which stated in electronic medical record
Arm/Group | AKI-RRT | AKI Non RRT
All-Cause Mortality (participants affected / at risk) | 96/302 | 34/811
Serious Adverse Events (participants affected / at risk) | 104/302 | 46/811
Other Adverse Events (participants affected / at risk) | 129/302 | 151/811
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKI-RRT (N=302) | AKI Non RRT (N=811)
Postoperative use of IABP (Cardiac disorders) | 104 | 46 — Sign of cardiac dysfunction that lead to the requirement of IABP
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKI-RRT (N=302) | AKI Non RRT (N=811)
Use of inotropes and vasoactive >2 drug (Vascular disorders) | 129 | 151 — Hemodynamic unstable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT06091982/Prot_SAP_000.pdf